CLINICAL TRIAL: NCT01224080
Title: Use of Adiana Tubal Occlusive Devices in Women With Hydrosalpinx Prior to In Vitro Fertilization
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reproductive Science Center (Industry)
Responsible Party: Donald Galen M.D., Reproductive Science Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVF-002
Record Dates: First submitted 2010-10-15; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Women Suffering From Unilateral or Bilateral Tubal Occlusion Due to Hydrosalpinx

ARMS (1):
- Adiana Device (Experimental): All patients will undergo the Adiana Tubal Occlusion procedure. This procedure will be done in an office based setting and last approximately 1 hour.
  Interventions: Device: Adiana placement

INTERVENTIONS:
Device: Adiana placement — All patients will undergo the Adiana Tubal Occlusion procedure. This procedure will be done in an office based setting and last approximately 1 hour.

SUMMARY:
A condition called hydrosalpinx occurs when one or both of the fallopian tubes is blocked with fluid. The fluid can leak into the tube and the uterus. The theory is that the fluid can harm the tubes and uterus making implantation more difficult or harm the embryo.

ELIGIBILITY:
Inclusion Criteria:

* Are willing to participate in this clinical study
* Are able to comprehend and give informed consent for participation in this study
* Have read, understood and signed an informed consent form
* Have been unable to achieve pregnancy after trying for 1 year or greater and who have unilateral or bilateral hydrosalpinges as evidenced by laparoscopy or ultrasound or HSG
* Have a Day #3 serum FSH<10, and Day #3 Estradiol<80
* Recipient women undergoing a ovum donor cycle the donor must have a Day 3 serum FSH < 10 and Day 3 Estradiol < 80
* Have an antral follicle count 10 or greater for both ovaries combined, if women using ovum donor (follicle count) will be based on eligible donor
* Have a desire to receive treatment for their HS
* Are willing to undergo a hysterosalpingogram (HSG) 3 months after ADIANA placement to confirm proximal tubal occlusion

Exclusion Criteria:

* Active or recent upper or lower pelvic infection
* Known hypersensitivity to nickel as confirmed by skin test
* Known allergy to contrast media
* Pregnancy or suspected pregnancy
* Delivery or termination of pregnancy less than six weeks prior to Adiana placements
* BMI > 35
* Abnormal pap smear (CIN2 or greater abnormality) within the past year
* Pelvic malignancy
* Severely retroverted uterus
* Evidence of intrauterine abnormalities such as submucous fibroids, polyps, intrauterine adhesions or presence of a uterine septum
* Abnormal Clomid Challenge Test or abnormal lab values on Day #3 serum FSH and Estradiol
* Antral follicle count less than 10 (both ovaries combined)
* Poor general or gynecologic health
* Inability or refusal to provide informed consent

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the success rate of proximal tubal occlusion with Adiana inserts in women with hydrosalpinx | 1 Year
  Analysis of results will be performed on the intent-to-treat population defined as all subjects in whom device placement was attempted and on the per protocol population defined as all subjects who had successful placement of the Adiana occlusion device and were followed for a minimum of one year post HSG confirmation test.

SECONDARY OUTCOMES:
Observe implantation and clinical pregnancy rates post IVF | 1Year
  Factors affecting the placement rate, tubal occlusion rate, and clinical pregnancy rate will be reviewed. This study employs an unblended, non randomized, single group design, in which subjects serve as their own controls. Because this feasibility study will enroll a maximum of ten (10) subjects, it is not designed with success/failure benchmarks, nor is it statistically powered to make any claims regarding effectiveness of hysteroscopic proximal tubal occlusion in women with hydrosalpinx who are planning to undergo IVF.

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Science Center, San Ramon, California, United States